CLINICAL TRIAL: NCT03382002
Title: Evaluation of Association Between Oxidative Parameters in Fertilization Medium of Cumulus Oocyte Complex (COC( as Measured by the TCL Assay and Clinical and Laboratory Outcome Parameters in IVF
Brief Title: Association Between Oxidative Parameters in Fertilization Medium of Cumulus Oocyte Complex and Outcome in IVF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Zofnat Wiener, Principal investigator, Carmel Medical Center
Other Study IDs: CarmelMC
Record Dates: First submitted 2017-11-29; First posted 2017-12-22 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Oxidative Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: TCL — evaluation of oxidative status

SUMMARY:
Medium of cumulus-oocyte complex will be assessed for oxidative status.

ELIGIBILITY:
Inclusion Criteria:

•Patients undergoing in vitro fertilization treatment

Exclusion Criteria:

•Patients undergoing intracytoplasmic sperm injection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female only
Study Population: Patients undergoing in vitro fertilization
Sampling Method: Non-Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-11-28 (Estimated); Study Completion 2020-04-28 (Estimated)

PRIMARY OUTCOMES:
Association of parameters of oxidative state with cycle outcome (pregnancy: yes/no) | two years
  The oxidative status in the incubation medium of the cumulus-oocyte complex will be assessed looking for an association between oxidative parameters and cycle outcome (pregnancy: yes/no))

CONTACTS AND LOCATIONS:
Locations (1):
- Carmel medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No